CLINICAL TRIAL: NCT06714617
Title: A Phase 1 Open-Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of BL-M17D1 in Subjects With HER2-Expressing or HER2-Mutant Advanced or Metastatic Solid Tumors
Brief Title: Evaluate BL-M17D1 in Patients w/HER2-Expressing/Mutant Advanced or Metastatic Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: SystImmune Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BL-M17D1-ST-101
Record Dates: First submitted 2024-11-27; First posted 2024-12-03 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer Stage III; HER2-positive Metastatic Breast Cancer; Unresectable Breast Carcinoma; Her2-Positive; HER2 Gene Mutation; Gastroesophageal-junction Cancer; Non Small Cell Lung Cancer; Endometrial Neoplasms; Peritoneal Cancer; Fallopian Tube Cancer; Ovarian Cancer; Urothelial Carcinoma Bladder; Solid Tumor, Adult; Gastric Cancer
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Endometrial Neoplasms; Fallopian Tube Neoplasms; Ovarian Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Escalation (Experimental): Beginning with Cycle 1, BL-M17D1 will be administered on Day 1 and Day 8 by (IV) infusion every 3 weeks (D1,D8 Q3W)
  Interventions: Drug: BL-M17D1
- Dose Finding (Experimental): Beginning with Cycle 1, BL-M17D1 will be administered on Day 1 and Day 8 by (IV) infusion every 3 weeks (D1,D8 Q3W)
  Interventions: Drug: BL-M17D1
- Dose Expansion (Experimental): Beginning with Cycle 1, BL-M17D1 will be administered on Day 1 and Day 8 by (IV) infusion every 3 weeks (D1,D8 Q3W)
  Interventions: Drug: BL-M17D1

INTERVENTIONS:
Drug: BL-M17D1 — The study includes 3 parts: Part 1 Dose escalation. Part 2 Dose Finding non-randomized and Part 3 Dose expansion randomized. BL-M17D1 will be administered on Day 1 and Day 8 by intravenous infusion every 3 weeks.

SUMMARY:
The objective of this study to evaluate the safety, tolerability, pharmacokinetics, and efficacy of BL-M17D1 in patients with HER2-Expressing or HER2-Mutant Advanced or Metastatic Solid Tumors.

DETAILED DESCRIPTION:
BL-M17D1-ST-101 is a multicenter, Phase 1 study evaluating the safety, tolerability, pharmacokinetic profile, and initial efficacy of BL-M17D1 in subjects with unresectable locally advanced or metastatic HER2-expressing or HER2-mutant solid tumors. This study will be conducted in three parts (dose escalation, dose finding and dose expansion). BL-M17D1 will be administered on Day 1 and Day 8 of a continuous 21-day treatment cycle.

ELIGIBILITY:
Inclusion Criteria:

1. Signed the informed consent form
2. Age ≥18 years.
3. Weighs more than 40 kg. For doses <0.3 mg/kg, subject must weigh ≥70 kg.
4. Has a life expectancy of ≥3 months.
5. Has documented locally advanced or metastatic HER2-positive solid tumor(s) (IHC 1+ to 3+ or in situ hybridization [ISH] positive) or HER2-mutant tumor specimen not amenable to curative surgery or radiation and has received at least 1 line of standard therapy in the advanced/metastatic setting, or for which no standard treatment is available, including:

   1. Cohort 1: HER2-positive breast cancer (BC);
   2. Cohort 2: HER2-positive gastric/gastroesophageal junction cancer (GC/GEJ);
   3. Cohort 3: HER2-positive or HER2-mutant non-small cell lung cancer (NSCLC);
   4. Cohort 4: HER2-positive endometrial cancer (EC);
   5. Cohort 5: HER2-positive ovarian cancer (OC), including fallopian tube cancer and primary peritoneal cancer;
   6. Cohort 6: HER2-positive urothelial cancers (UC);
   7. Cohort 7: Other HER2-positive solid tumors as approved by the medical monitor. Note: For indications in which a HER2-directed therapy is approved, the approved treatment is recommended although not mandated, at the discretion of the investigator.
6. Agree to provide most recent existing tumor samples (FFPE tissue block or slides) from primary or metastatic sites for tissue-based IHC staining to centrally determine HER2 expression:

   1. In dose escalation and dose finding: archival tissue or fresh biopsy. If no archival tissue is available or it is not possible to obtain a fresh tissue biopsy, medical monitor approval is required;
   2. In dose expansion: an FFPE block or slides from fresh biopsy or the most recent archival tissue is required.
7. Has at least one measurable lesion based on RECIST (Response Evaluation Criteria in Solid Tumors) V1.1.
8. Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 to 1.
9. Toxicity of previous antitumor therapy has returned to Grade ≤1 as defined by NCI CTCAE V5.0, except for alopecia and endocrinopathies controlled by replacement therapy that must be Grade ≤2.
10. No serious cardiac dysfunction and left ventricular ejection fraction ≥50%.
11. Has adequate organ function before enrollment, defined as:

    1. Marrow function: Absolute neutrophil count (ANC) ≥1.5×109/L, platelet count ≥100×109/L, hemoglobin (Hb) ≥9.0 g/dL (blood transfusion, platelet transfusion, erythropoietin, platelet-stimulating agents, and G-CSF use are not allowed 1 week prior to screening);
    2. Hepatic function: Total bilirubin (TBIL) ≤1.5×ULN (≤3×ULN for subjects with Gilbert's syndrome or liver metastasis at baseline), AST and ALT without liver metastasis ≤3.0×ULN, AST and ALT with liver metastasis ≤5.0×ULN;
    3. Renal function: Creatinine (Cr) clearance ≥60 mL/minute (Cockcroft-Gault equation).
12. Coagulation parameters: International normalized ratio (INR) ≤1.5×ULN, and activated partial thromboplastin time (aPTT) ≤1.5×ULN, unless receiving anticoagulation therapy with PT and aPTT levels within the intended therapeutic range.
13. Urine protein ≤2+ or ≤1000 mg/24 hours.
14. Sexually active fertile subjects and their partners must agree to use highly effective methods of contraception during the course of the study and for 7 months after the last dose of study treatment. An additional contraceptive method, such as a barrier method (eg, condom), is recommended.
15. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test at screening and must be nonlactating. Female subjects are considered WOCBP unless one of the following criteria are met: documented permanent sterilization (hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) or documented postmenopausal status (defined as 12 months of amenorrhea in a woman >45 years old in the absence of other biological or physiological causes. In addition, females <55 years old must have a serum follicle stimulating hormone (FSH) level >40 mIU/mL to confirm menopause.

Note: Documentation may include review of medical records, medical examination, or medical history interview by study site staff.

Exclusion Criteria:

Subjects who meet any of the following criteria will not be eligible for participation in this study:

1. Chemotherapy, biological therapy, immunotherapy, radical radiotherapy, targeted therapy (including small molecule inhibitor of tyrosine kinase), and other antitumor therapy within 4 weeks or 5 half-lives (whichever is shorter) prior to the first administration; major surgery within 4 weeks prior to the first administration; mitomycin and nitrosoureas treatment within 6 weeks prior to the first administration.
2. Concomitant use of strong inhibitors and inducers of any CYP3A4 enzyme or P-gp transporter system within 2 weeks or 5 half-lives (whichever is longer) prior to the first administration and throughout all parts of the study.
3. History of severe heart disease, such as symptomatic congestive heart failure (CHF) ≥ Grade 2 (CTCAE 5.0), New York Heart Association (NYHA) ≥ Grade 2 heart failure at any time, or history of myocardial infarction or unstable angina pectoris within 6 months before enrollment.
4. Prolonged QT interval (QTcF >470 msec), complete left bundle branch block, Grade 3 atrioventricular block, or a history of additional risk factors for torsades de pointes (TdP; eg, heart failure as defined in Exclusion Criterion 3, chronic or recurrent hypokalemia that requires medical intervention, congenital long QT syndrome, family history of long QT syndrome) or any current concomitant medication known to prolong the QT/QTc interval or cause TdP.
5. Active autoimmune diseases and inflammatory diseases, such as systemic lupus erythematosus, psoriasis requiring systemic treatment, rheumatoid arthritis, inflammatory bowel disease and Hashimoto's thyroiditis, etc., except for type 1 diabetes, hypothyroidism that can be controlled by standard of care treatment, and skin diseases that do not require systemic treatment (such as vitiligo, psoriasis).
6. Other prior malignancies except for basal cell carcinoma of the skin, squamous cell carcinoma of the skin and/or carcinoma in situ after adequate resection, or other malignancy treated with curative intent with a disease-free interval of at least 3 years prior to screening.
7. Poorly controlled hypertension by two types of antihypertensive drugs (systolic blood pressure >150 mmHg or diastolic blood pressure >100 mmHg).
8. Advanced or clinically significant lung diseases, such as poorly controlled chronic obstructive pulmonary disease and asthma, restrictive lung disease, pulmonary hypertension etc.
9. Have a history of noninfectious interstitial lung disease (ILD)/pneumonitis that required treatment with steroids, have current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening.
10. Stroke or transient ischemic attack (TIA) within 6 months before enrollment.
11. Thromboembolic event (eg, deep vein thrombosis [DVT] or pulmonary embolism [PE]) within 6 months before enrollment except for those who are clinically stable and receiving treatment with adequate anticoagulant therapy for at least 3 weeks before enrollment.
12. Primary tumors in the central nervous system (CNS) and active or untreated CNS metastases and/or carcinomatous meningitis should be excluded. Patients with previously treated brain metastases may participate provided they are clinically stable for at least 4 weeks and have no evidence of new or enlarging brain metastases and no requirements for corticosteroids 14 days prior to dosing with the IP. Patients on low dose corticosteroids (<10 mg prednisone or equivalent/day) may participate.
13. Pre-existing ≥Grade 2 peripheral neuropathy.
14. Subjects who have a history of anaphylaxis or severe hypersensitivity to recombinant humanized antibodies or human-mouse chimeric antibodies or any of the components of BL-M17D1.
15. Subjects who are receiving treatment with systemic glucocorticoids >10 mg/day equivalent of prednisone, except for the treatment of chronic obstructive pulmonary disease, antiemetic, infusion reactions; however, treatment with low dose glucocorticoids (≤10 mg/day equivalent of prednisone) is permitted. The chronic use of topical, inhaled, and locally injected steroids is permitted.
16. Known human immunodeficiency virus (HIV) infection (HIV antibody positive). Subjects are allowed to participate if all the following criteria are met:

    1. Undetectable HIV RNA and CD4 count ≥ 350 cells/μL at screening;
    2. No AIDS-defining opportunistic infection within 12 months prior to screening;
    3. On stable antiretroviral therapy (ART) for at least 4 weeks prior to enrollment with projected continuation of ART as clinically indicated while on the study.
17. Active hepatitis B virus (HBV) infection (positive HBsAg test). Subjects with a chronic inactive HBV infection are eligible if all the following criteria are met:

    1. HBV DNA viral load < 500 IU/mL;
    2. Normal AST and ALT, OR if liver metastasis is present, have AST and ALT <3×ULN which are not attributed to HBV infection;
    3. Are on antiviral treatment, as clinically indicated.
18. Active hepatitis C virus (HCV) infection (HCV antibody positive and HCV RNA > the lower limit of detection). Subjects with a positive anti-HCV antibody are eligible only if PCR is negative for HCV RNA.
19. Active or latent tuberculosis.
20. Active infections requiring IV antibiotic, antiviral, or antifungal treatment, such as severe pneumonia, bacteremia, sepsis, etc., within 1 week prior to first dose of study treatment. Subjects on stable oral antimicrobials with no clinical or laboratory evidence of active infection are eligible.
21. Participated in another clinical trial within 4 weeks prior to first dose of study treatment.
22. Pregnant, breastfeeding, or planning to become pregnant during the study.
23. Other conditions that the investigator or sponsor believes are not suitable for participating in this clinical trial.
24. Received prior treatment with an ADC with a microtubule inhibitor payload.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Participants with Dose-limiting toxicities | 1 Year
  Measuring the number of patients Dose-limiting toxicities (DLTs). A DLT is defined as any of the following events that are not clearly due to the underlying disease or extraneous causes:
  Hematologic toxicities
  * Grade 4 neutrophil count decreased lasting >7 days
  * Grade ≥3 febrile neutropenia of any duration
  * Grade ≥3 platelet count decreased with clinically significant hemorrhage
  * Grade 4 thrombocytopenia lasting >7 days Nonhematologic toxicities
  * Death not clearly related to disease progression or extraneous cause
  * Hy's law cases
  * Grade ≥3 nonhematologic toxicities
Participants with Serious Adverse Events (SAEs) and treatment-emergent adverse events (TEAEs) | 1 Year
  Measuring the number of patients with serious adverse events (SAEs) and treatment-emergent adverse events (TEAEs)
To determine the MTD if reached or MAD and two or more RDEs of BL-M17D1 | 1 Year
  MTD, MAD, and RDE

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Tannenbaum, MD, MSc, Study Chair — SystImmune Inc.
Locations (9):
- United States (9):
  - SCRI-Denver HealthOne, Denver, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - SCRI-Florida Cancer Center Specialists Lake Mary, Lake Mary, Florida
  - Hematology Oncology Associates of the Treasure Cost, Port Saint Lucie, Florida
  - SCRI-Florida Cancer Center Specialists Sarasota, Sarasota, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - SCRI-Sidney Kimmel Cancer Center, Philadelphia, Pennsylvania
  - SCRI-Oncology Partners, Nashville, Tennessee
  - NEXT Oncology, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No